CLINICAL TRIAL: NCT02412176
Title: A Comparison Between Right Ventricular Apical Pacing and True Mid-septal Pacing, Verified With Computed Tomography: a Randomized Study
Brief Title: Right Ventricular Apical Versus True Mid-septal Pacing
Acronym: MS-R
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Pavel Osmancik, Charles University in Prague, Czech Republic, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CharlesUCR
Record Dates: First submitted 2015-03-24; First posted 2015-04-09 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Ventricular Rhythm From Artificial Pacing
Keywords: pacemaker; dyssynchrony; apical pacing; mid-septum
MeSH Terms: interventions — Deoxyribonuclease (Pyrimidine Dimer)

STUDY DESIGN:
Intervention Model Description: RV lead in the apex
Who Masked: Participant
Masking Description: RV lead in the septum
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pacing site - right ventricular apex (Experimental): The intervention will be the implantation of the lead into the right ventricular apex
  Interventions: Procedure: Pacing site - the implantation in the right ventricular (RV) apex
- Pacing site - septum (Experimental): The intervention will be the implantation of the lead into the septum.
  Interventions: Procedure: Pacing site - the implantation in the septum

INTERVENTIONS:
Procedure: Pacing site - the implantation in the right ventricular (RV) apex — Pacing site - RV apex. The lead will be implanted in the RV apex.
  Other Names: Pacing site - RV apex
  Arms: Pacing site - right ventricular apex
Procedure: Pacing site - the implantation in the septum — Pacing site - septum. The lead will be implanted in the septum.
  Other Names: Pacing site - MS
  Arms: Pacing site - septum

SUMMARY:
Background Right ventricular (RV) artificial apical pacing can negatively impact synchrony of left ventricular contraction. The pacing from the septum of the RV can present an advantage in terms of less expressed dyssynchrony and reduced negative impact on left ventricular (LV) function. However, results of randomized studies comparing apical and septal pacing are not uniform. All these results have been affected by improper implantation of the septal lead, with many apparently septal leads being, in fact, implanted off-septum. The aim of the study is to compare true septal pacing with other RV pacing locations.

Methods/Design This is a prospective, randomized, single center study. Patients with standard indications for cardiac pacing with the expectation of high percentage RV pacing will be enrolled. They will be randomized into apical and septal pacing. The real location of leads in patients randomized to septal pacing will be confirmed using cardiac CT. After cardiac CT, three groups of patients will be created: 1) apical pacing, 2) true septal (in which the position of the lead has been verified to be in the septum), and 3) apparent septal (in which the position of the lead was found to be off-septum). Primary end-point are changes in standard echocardiographic parameters (LV ejection fraction, LV end-systolic volume, and LV end-diastolic volume) and the concentration of N-terminal pro brain natriuretic peptide (NT-proBNP) from baseline to 6 months, 1 year and three years. Secondary end-points are changes in echo-parameters of LV synchrony.

Discussion It is hypothesized that correct septal pacing will be associated with reduce negative impact on the function of the left ventricle (i.e. smaller decreases in LV EF and smaller increases in LVEDV, LVESV) and NT-proBNP, and less expressed LV dyssynchrony.

DETAILED DESCRIPTION:
METHODS/DESIGN The study is planned as prospective, multicenter, randomized study. The study was approved by the local ethics committee, and written informed consent will be obtained before enrollment of patients.

Inclusion criteria will be the following:

1. Indication for cardiac pacing based on recent guidelines of European Society of Cardiology (5)
2. High degree atrio-ventricular (AV) block (AV block 2/1 or second degree AV block with resulting heart rate below 50), or atrial fibrillation with slow conduction to ventricles.
3. A high probability of needing significant ventricular stimulation (more than 50%)
4. Written informed consent.

Exclusion criteria will be the following:

1. The absence of written informed consent
2. Renal insufficiency (creatinine level more than 130 µmol/l)
3. History of Iodine allergy
4. Claustrophobia
5. Significant valve disease (i.e. mitral insufficiency 75% and worse, moderate or severe aortic stenosis)
6. Recent (within three months) acute coronary syndrome
7. Planned cardiac surgery (coronary artery bypass grafting, valve surgery)
8. Ejection fraction of left ventricle less than 50%
9. Expected life expectancy less than 3 years
10. Expected non-compliance.

End-points: there are three unique primary end-points: 1) changes in left ventricular end-systolic volume (LVESV) over time (from baseline to 6 months and 3 years), 2) changes in the left ventricular ejection fraction (LV EF) over time (from baseline to 6 months and 3 years) and 3) changes in concentration of N-terminal pro brain natriuretic peptide (NT-proBNP), from baseline to 6 months up to three years).

Secondary endpoints are changes in echocardiography parameters of left ventricular synchrony, changes in left ventricular end-diastolic volume (LVEDV) over time and changes in the quality of life, as assessed by the Minnesota Living with Heart Failure questionnaire, over time (from baseline to 6 months and 3 years).

Power calculation and statistical analysis: The sample size calculation was based on the following assumptions: the power of the test = 0.8 and a statistical significance border = 0.05. Based on information from previous trials regarding the effect of pacing on left ventricular volumes and parameters, it is assumed that there will be at least a 10% difference in the change of LV end-systolic volume (LVESV, measured from baseline to 3 years follow-up) between the group paced from apex and the group with true septal pacing. Based on previous results regarding the efficacy of true septal pacing, based on recent fluoroscopy criteria, it is assumed that approximately 40% of those randomized to the septal group will not have the lead located in the septum, but in the anterior wall. This means that 70 patients are needed in the apical group, 70 in the septal group and 70 in the apparent septal group to achieve statistical significance. Data analysis will be performed using standard tests (chi-square, Student t-test, Kruskal-Wallis test etc.) For data description, standard descriptive statistical methods will be used: absolute and relative frequencies for categorical data and the median with 5-95% percentiles for continuous data. For categorical variables, statistical analysis will be done using the χ2 or the Fisher exact test; for continuous variables, the Student t-test, Mann-Whitney U test or Kruskal-Wallis test will be used. Kaplan-Meier curves will be calculated for visualizing the occurrence of end-points during follow-up. The influence of patient characteristics on the occurrence of end-points will be calculated using logistic regression and the Cox proportional risk model, when appropriate.

Data analysis In the primary analysis, three groups of patients will be analyzed: 1) patients randomized to RV apical pacing (apex group); 2) patients with true septal pacing (true septal group, i.e. those randomized to septal pacing, in whom the location of the lead was confirmed (using cardiac CT) to actually be in the septum), and 3) patients with apparent septal pacing (apparent septal group, i.e. those randomized to septal pacing, in whom the lead location will be found to off-septum, based on cardiac CT). The primary goal of the study will be to confirm that true septal pacing is associated with fewer prominent negative effects on the left ventricle. A secondary goal is to determine if off-septum placement (i.e., apparent septal group) has similar negative consequences for the left ventricle as those seen in apical pacing. In a secondary analysis, the two original groups will be compared (i.e., the groups randomized to apical vs. septal pacing).

Echocardiographic evaluation All patients will undergo echocardiography before implantation and during follow-up. Echocardiography will be done in the left lateral decubitus position. Imaging will be performed using a commercially available echocardiographic system (VIVID 7, General Electric Ultrasound, Milwaukee, USA). Images will be obtained using a 3.5 Mega Hertz transducer, at a depth of 16 cm in the parasternal (long and short axis) and apical (two- and four-chamber images) views. Standard 2D and colour Doppler data, triggered by the Q R S complex, will be saved in cine-loop format. A minimum of three consecutive beats will be recorded from each view and the images will be digitally stored for off-line analysis (EchoPac 7.0.0, General Electric Ultrasound, Milwaukee, USA). Left ventricular end-systolic volume (LVESV), LV end-diastolic volume (LVEDV), and LV EF will be measured from the apical two- and four-chamber images, using the (modified biplane) Simpson's rule. (10) Parameters of interventricular and left ventricular dyssynchrony will be measured off-line using tissue Doppler.

Conventional tissue Doppler-based dyssynchrony indices will be determined; (11) the standard deviation (SD) in time to peak velocity in 12 mid and basal segments (Ts SD12), the difference in time to peak velocity between anteroseptal and posterior wall (Ts AsP), the difference in time to peak velocity between the septal and lateral wall (Ts SL) as well as the maximal difference in time to peak velocity in 6 basal segments (Ts Diff6). Moreover, newer recently published parameters of dyssynchrony, such as apical rocking or septal flash, will also be measured. (12)

Further examinations before implantation Patients will be asked to complete the Minnesota Living with Heart Failure Questionnaire and the concentration of NT-proBNP, in peripheral blood will be measured. Afterwards patients will be randomized to RV apical or RV septal pacing. Because it can be anticipated that not all leads intended for RV septal implantation will actually end up implanted in the RV septum (some will be in the free anterior wall or in the anteroseptal groove), the ratio of randomization will be 2/1 (mid-septal vs. apical).

Implantation will be done using the standard approach, i.e., using the subclavian or cephalic approach. Only active fixation leads will be used. The position of the lead in the RV apical group will be assessed by displaying the lead in the anteroposterior (AP), right anterior oblique (RAO) 30 and left anterior oblique (LAO) 40 projection and stored. For the septal pacing group, a 3D stylet with two angulations will be prepared, as proposed recently. (9) Initially, the distal end of a standard stylet will be manually shaped into a smooth large curve, in a single plane, over a length of about 20 cm using the barrel of a syringe. The lead, with this J-shape stylet, will be advanced into the RV and further to the pulmonary artery. Then the stylet will be withdrawn and an additional 90° curve angulation will be created with the distal 3 cm end of the stylet. The 3D stylet will be inserted into the lead, and by slight counterclockwise torque applied, the lead will be withdrawn from the pulmonary artery to the right ventricle. A "jump" is usually seen as the lead falls below the RV outflow tract. At that point, the lead is quickly advanced and forced against the mid-septum. This manipulation will be done using RAO 30, and the target position is in the middle of the cardiac contour. Before final lead fixation, the position of the lead will be checked in the LAO 40 (the lead should point toward the spine with an angle to the horizontal plane between 0 to 60°). Perioperative fluoroscopy images will be stored, and standard implant parameters will be measured (impedance, R wave amplitude, and threshold).

Cardiac CT will be performed 6-12 weeks after implantation to assess the true position of the RV lead in the heart. Before cardiac CT, lead dislodgement will be excluded by measuring standard lead parameters.

Image acquisition CT will be performed using a 256-detector-row CT scanner (Brilliance CT 256; Philips, Best, The Netherlands) with a tube voltage of 100 kilo Volt (kV), collimation of 2x128×0.625 mm, a pitch of 0.18, a rotation time of 0.27 s, and a slice thickness of 0.9 mm. A tri-phasic injection of 60 mL of contrast media (Ultravist 370, Bayer Healthcare Pharmaceuticals, New Jersey, USA) will be used. Initially, 50 mL of contrast agent will be administered at a flow rate of 4.0 mL/s, followed by 20 mL of 50% contrast/saline. Subsequently, a saline flush of 30 mL will be administered at a flow rate of 3.0 mL/s. Bolus tracking will be used for synchronization of the contrast medium injection during scanning. The region of interest will be the descending aorta. After enhancement reaches 140 hounsfield Units (HU), there will be 3-s post-threshold delay before the scan is commenced. Prospective ECG triggered dose modulation (mode "step and shoot") will be used, scanning 70-80% of the R - R interval. After examination, the displayed dose-length product (DLP) will be recorded to evaluate radiation dose.

Image post-processing Datasets will be transferred to an external workstation (Comprehensive Cardiac Analyses, Brilliance Workspace v 4.0, Philips Healthcare, Cleveland, USA) for off-line analysis. Axial slices, oblique reconstructions and maximum-intensity projection (MIP) images will be used for precise localization of the RV lead. According to the location of RV lead, septal group patients will be divided in two sub-groups: true septum group (i.e. patients randomize to septal pacing, in whom the lead is actually found to be in the septum) and apparent septum group (i.e. those randomized to the septal pacing, in whom the lead is found to be off-septum, and typically in the free anterior wall or in the anteroseptal groove). Because the apical position is easily visible with fluoroscopy, cardiac CT will be done only in the patients randomized to septal pacing.

Post-implantation follow-up and out-patient controls will be done at 6 months, 1 year, and 3 years. During each control, standard pacemaker parameters (impedance, threshold, and amplitude) will be measured, and the percentage of ventricular stimulation will be assessed. During each control, echocardiography will be done, NT-proBNP measured, and patients will be asked to fulfill the Minnesota questionnaire.

ELIGIBILITY:
Inclusion Criteria:

Indication for cardiac pacing.

Exclusion Criteria:

* renal insufficiency
* iod allergy
* claustrophobia
* significant valvular disease
* recent acute coronary syndrome
* planned cardiac surgery
* ejection fraction of left ventricle less than 50%
* live expectancy less than 3 years
* expected non-compliance of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the left ventricular ejection fraction at 6 months | from baseline to 6 months
  The changes over time in the left ventricular ejection fraction will be determined.
Change from baseline in the left ventricular end-systolic volume at 6 months | from baseline to 6 months
  The changes over time in the left ventricular end-systolic volume will be determined.
Change from baseline in the concentration of N-terminal pro-Brain Natriuretic Peptide at 6 months | from baseline to 6 months
  The changes over time in the concentration of the N-terminal pro-brain natriuretic peptide will be determined.
Change from baseline in the left ventricular ejection fraction at 3 years | from baseline to 3 years
  The changes over time in the left ventricular ejection fraction will be determined.
Change from baseline in the left ventricular end-systolic volume at 3 years. | from baseline to 3 years
  The changes over time in the left ventricular ejection fraction will be determined.
Change from baseline in the concentration of N-terminal pro-Brain Natriuretic Peptide at 3 years. | from baseline to 3 years
  The changes over time in the concentration of the N-terminal pro-brain natriuretic peptide will be determined.

SECONDARY OUTCOMES:
Change from baseline in dyssynchrony at 6 months | from baseline to 6 months
  Echo parameters of dyssynchrony wil be measured.
Change from baseline in the left ventricular end-diastolic volume at 6 months | from baseline to 6 months
  The changes over time in the left ventricular end-diastolic volume will be determined.
Change from baseline in dyssynchrony at 3 years. | from baseline to 3 years
  Echo parameters of dyssynchrony wil be measured.
Change from baseline in the left ventricular end-diastolic volume at 3 years. | from baseline to 3 years
  The changes over time in the left ventricular end-diastolic volume will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Osmancik, MD, PhD, Principal Investigator — 3rd Faculty of Medicine, Charles University Prague
Locations (1):
- Charles University in Prague, Prague, Czechia

REFERENCES:
- [Background] Burri H, Domenichini G, Sunthorn H, Ganiere V, Stettler C. Comparison of tools and techniques for implanting pacemaker leads on the ventricular mid-septum. Europace. 2012 Jun;14(6):847-52. doi: 10.1093/europace/eur404. Epub 2011 Dec 26. PMID 22201018
- [Background] Curtis AB, Worley SJ, Adamson PB, Chung ES, Niazi I, Sherfesee L, Shinn T, Sutton MS; Biventricular versus Right Ventricular Pacing in Heart Failure Patients with Atrioventricular Block (BLOCK HF) Trial Investigators. Biventricular pacing for atrioventricular block and systolic dysfunction. N Engl J Med. 2013 Apr 25;368(17):1585-93. doi: 10.1056/NEJMoa1210356. PMID 23614585
- [Result] Tse HF, Lau CP. Long-term effect of right ventricular pacing on myocardial perfusion and function. J Am Coll Cardiol. 1997 Mar 15;29(4):744-9. doi: 10.1016/s0735-1097(96)00586-4. PMID 9091519
- [Result] Zhang XH, Chen H, Siu CW, Yiu KH, Chan WS, Lee KL, Chan HW, Lee SW, Fu GS, Lau CP, Tse HF. New-onset heart failure after permanent right ventricular apical pacing in patients with acquired high-grade atrioventricular block and normal left ventricular function. J Cardiovasc Electrophysiol. 2008 Feb;19(2):136-41. doi: 10.1111/j.1540-8167.2007.01014.x. Epub 2007 Nov 12. PMID 18005026
- [Result] Shimony A, Eisenberg MJ, Filion KB, Amit G. Beneficial effects of right ventricular non-apical vs. apical pacing: a systematic review and meta-analysis of randomized-controlled trials. Europace. 2012 Jan;14(1):81-91. doi: 10.1093/europace/eur240. Epub 2011 Jul 27. PMID 21798880
- [Result] Domenichini G, Sunthorn H, Fleury E, Foulkes H, Stettler C, Burri H. Pacing of the interventricular septum versus the right ventricular apex: a prospective, randomized study. Eur J Intern Med. 2012 Oct;23(7):621-7. doi: 10.1016/j.ejim.2012.03.012. Epub 2012 Apr 11. PMID 22939807
- [Result] Vardas PE, Auricchio A, Blanc JJ, Daubert JC, Drexler H, Ector H, Gasparini M, Linde C, Morgado FB, Oto A, Sutton R, Trusz-Gluza M; European Society of Cardiology; European Heart Rhythm Association. Guidelines for cardiac pacing and cardiac resynchronization therapy: The Task Force for Cardiac Pacing and Cardiac Resynchronization Therapy of the European Society of Cardiology. Developed in collaboration with the European Heart Rhythm Association. Eur Heart J. 2007 Sep;28(18):2256-95. doi: 10.1093/eurheartj/ehm305. Epub 2007 Aug 28. No abstract available. PMID 17726042
- [Result] Burri H, Park CI, Zimmermann M, Gentil-Baron P, Stettler C, Sunthorn H, Domenichini G, Shah D. Utility of the surface electrocardiogram for confirming right ventricular septal pacing: validation using electroanatomical mapping. Europace. 2011 Jan;13(1):82-6. doi: 10.1093/europace/euq332. Epub 2010 Sep 9. PMID 20829188
- [Result] Osmancik P, Stros P, Herman D, Curila K, Petr R. The insufficiency of left anterior oblique and the usefulness of right anterior oblique projection for correct localization of a computed tomography-verified right ventricular lead into the midseptum. Circ Arrhythm Electrophysiol. 2013 Aug;6(4):719-25. doi: 10.1161/CIRCEP.113.000232. Epub 2013 Jun 6. PMID 23742805
- [Result] Schiller NB, Shah PM, Crawford M, DeMaria A, Devereux R, Feigenbaum H, Gutgesell H, Reichek N, Sahn D, Schnittger I, et al. Recommendations for quantitation of the left ventricle by two-dimensional echocardiography. American Society of Echocardiography Committee on Standards, Subcommittee on Quantitation of Two-Dimensional Echocardiograms. J Am Soc Echocardiogr. 1989 Sep-Oct;2(5):358-67. doi: 10.1016/s0894-7317(89)80014-8. PMID 2698218
- [Result] Yu CM, Zhang Q, Fung JW, Chan HC, Chan YS, Yip GW, Kong SL, Lin H, Zhang Y, Sanderson JE. A novel tool to assess systolic asynchrony and identify responders of cardiac resynchronization therapy by tissue synchronization imaging. J Am Coll Cardiol. 2005 Mar 1;45(5):677-84. doi: 10.1016/j.jacc.2004.12.003. PMID 15734610
- [Result] Szulik M, Tillekaerts M, Vangeel V, Ganame J, Willems R, Lenarczyk R, Rademakers F, Kalarus Z, Kukulski T, Voigt JU. Assessment of apical rocking: a new, integrative approach for selection of candidates for cardiac resynchronization therapy. Eur J Echocardiogr. 2010 Dec;11(10):863-9. doi: 10.1093/ejechocard/jeq081. Epub 2010 Jul 7. PMID 20615904
- [Result] Stockburger M, Gomez-Doblas JJ, Lamas G, Alzueta J, Fernandez-Lozano I, Cobo E, Wiegand U, Concha JF, Navarro X, Navarro-Lopez F, de Teresa E. Preventing ventricular dysfunction in pacemaker patients without advanced heart failure: results from a multicentre international randomized trial (PREVENT-HF). Eur J Heart Fail. 2011 Jun;13(6):633-41. doi: 10.1093/eurjhf/hfr041. PMID 21613427
- [Result] Padeletti L, Lieberman R, Schreuder J, Michelucci A, Collella A, Pieragnoli P, Ricciardi G, Eastman W, Valsecchi S, Hettrick DA. Acute effects of His bundle pacing versus left ventricular and right ventricular pacing on left ventricular function. Am J Cardiol. 2007 Nov 15;100(10):1556-60. doi: 10.1016/j.amjcard.2007.06.055. PMID 17996519
- [Result] Peschar M, de Swart H, Michels KJ, Reneman RS, Prinzen FW. Left ventricular septal and apex pacing for optimal pump function in canine hearts. J Am Coll Cardiol. 2003 Apr 2;41(7):1218-26. doi: 10.1016/s0735-1097(03)00091-3. PMID 12679225
- [Result] Vancura V, Wichterle D, Melenovsky V, Kautzner J. Assessment of optimal right ventricular pacing site using invasive measurement of left ventricular systolic and diastolic function. Europace. 2013 Oct;15(10):1482-90. doi: 10.1093/europace/eut068. Epub 2013 Apr 12. PMID 23585254
- [Result] Ng AC, Allman C, Vidaic J, Tie H, Hopkins AP, Leung DY. Long-term impact of right ventricular septal versus apical pacing on left ventricular synchrony and function in patients with second- or third-degree heart block. Am J Cardiol. 2009 Apr 15;103(8):1096-101. doi: 10.1016/j.amjcard.2008.12.029. Epub 2009 Feb 21. PMID 19361596
- [Derived] Mala A, Osmancik P, Herman D, Curila K, Stros P, Vesela J, Prochazkova R, Petr R. Can QRS morphology be used to differentiate between true septal vs. apparently septal lead placement? An analysis of ECG of real mid-septal, apparent mid-septal, and apical pacing. Eur Heart J Suppl. 2020 Jul;22(Suppl F):F14-F22. doi: 10.1093/eurheartj/suaa094. Epub 2020 Jul 15. PMID 32694949